CLINICAL TRIAL: NCT00531856
Title: A Prospective, Multicenter, Single-blind, Placebo-controlled, Safety and Tolerability Study of the Effects of Carbon Monoxide for Inhalation in Patients Receiving Kidney Transplants.
Brief Title: Safety and Tolerability Study of Inhaled Carbon Monoxide in Kidney Transplant Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical Hold pending additional data review and protocol amendment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C201
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplant, Carbon Monoxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 5.97 mg/L of carbon monoxide in 30% oxygen
  Interventions: Drug: Inhaled carbon monoxide
- 2 (Placebo Comparator): Oxygen 30% in Nitrogen
  Interventions: Drug: Inhaled carbon monoxide

INTERVENTIONS:
Drug: Inhaled carbon monoxide — 0.7 mg/kg carbon monoxide/placebo over one hour administered 12-48 hours post transplant
Drug: Inhaled carbon monoxide — 2.0 mg/kg carbon monoxide/placebo over one hour administered 12-48 hours post transplant
Drug: Inhaled carbon monoxide — 3.0 mg/kg carbon monoxide/placebo over one hour administered 12-48 hours during transplant
Drug: Inhaled Carbon Monoxide — 3.5 mg/kg carbon monoxide/placebo over one hour administered 12-48 hours during transplant
Drug: Inhaled Carbon Monoxide — 2.0 mg/kg carbon monoxide/placebo over one hour administered 12-48 hours during transplant.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of two carbon monoxide doses when administered as an inhaled gas for 1 hour in patients receiving kidney transplants.

DETAILED DESCRIPTION:
The mechanisms by which carbon monoxide exerts its effects in preventing damage of the graft appear to vary among the models and organs with the common theme of carbon monoxide acting as a potent anti-inflammatory molecule. Carbon monoxide affects several intracellular signaling pathways. In addition, carbon monoxide generates increased levels of anti-inflammatory molecules.

Evaluate the safety and tolerability of three carbon monoxide dose levels consisting of a single 0.7 mg/kg dose and a single 2.0 mg/kg dose when administered post-operatively and a single 2.0 mg/kg dose, a single 3.0mg/kg dose and a 3.5 mg/kg dose when administered intra-operatively as an inhaled gas for 1 hour, by assessment of adverse events (AEs), vital signs, laboratory variables, serum carboxyhemoglobin (COHb), oxygenation, electrocardiography (ECG), and neurocognitive status in patients receiving kidney transplants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female receiving a kidney transplant from any donor type
* BMI between 16 and 36 inclusive
* Spontaneously breathing (non-intubated) with supplemental oxygen standardized at 2 liters via nasal cannula
* Hemodynamically stable with a systolic arterial pressure > 90 mmHg and a heart rate < 120 beats/min
* Acceptable transplantation candidate as judged by medical history, physical exam, ECG, vital signs, clinical chemistry, hematology, and urinalysis
* Given written and verbal information and had the opportunity to ask questions about the study
* Signed informed consent to participate in the study

Exclusion Criteria:

* Exposure to any carbon monoxide source (e.g., fire, gas, or heavily polluted air) during the 48 hours prior to the study day
* Baseline blood level of COHb >2%
* Baseline hemoglobin (Hb) <10.0 g/dL
* Patients with significant underlying lung disease such as moderate or severe asthma, COPD, and interstitial lung disease
* Baseline oxygen saturation <95%
* Pregnancy or breastfeeding
* Participation in other clinical trial within 2 months prior to study drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of three carbon monoxide dose levels when administered as an inhaled gas for 1 hour in patients receiving kidney transplants | 28 days

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of the inhaled carbon monoxide; Correlate the safety parameters to inhaled carbon monoxide and COHb levels; Assess laboratory values; Assess potential markers for the incidence of delayed graft function | 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Universtiy of CA, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts